CLINICAL TRIAL: NCT07128550
Title: A Phase 3 Randomized, Open-Label Study to Evaluate the Efficacy and Safety of Tobevibart+Elebsiran Combination Therapy in Participants With Chronic HDV Infection Not Virologically Suppressed With Bulevirtide (ECLIPSE 2)
Brief Title: A Study to Evaluate Tobevibart+Elebsiran in Participants With Chronic HDV Infection Not Virologically Suppressed With Bulevirtide
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIR-CHDV-V205
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Viral Hepatitis
Keywords: HDV; Hepatitis D Virus; Hepatitis; Chronic Hepatitis D Virus; Hepatitis D; Hepatitis D, Chronic; Hepatitis Delta Virus; Digestive System Diseases; Liver Diseases
MeSH Terms: conditions — Hepatitis; Hepatitis D; Hepatitis D, Chronic; Digestive System Diseases; Liver Diseases | interventions — bulevirtide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants will receive treatment with tobevibart + elebsiran up to 240 weeks.
  Interventions: Drug: Tobevibart; Drug: Elebsiran
- Arm 2 (Experimental): Participants will receive Bulevirtide for 24 weeks and switch to receive tobevibart + elebsiran for additional 216 weeks
  Interventions: Drug: Tobevibart; Drug: Elebsiran; Drug: Bulevirtide

INTERVENTIONS:
Drug: Tobevibart — Tobevibart administered by subcutaneous injection
  Other Names: VIR-3434
Drug: Elebsiran — Elebsiran administered by subcutaneous injection
  Other Names: VIR-2218
Drug: Bulevirtide — Bulevirtide administered by subcutaneous injection
  Other Names: Hepcludex
  Arms: Arm 2

SUMMARY:
This is a multicenter, open label, randomized Phase 3 clinical study to evaluate tobevibart + elebsiran in participants with Chronic HDV Infection not virologically suppressed with bulevirtide

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages 18 to 70 years at screening
2. HDV RNA ≥ 500 IU/mL at screening
3. Receiving BLV 2 mg SC QD for ≥ 24 weeks at Day 1
4. Noncirrhotic or compensated cirrhotic liver disease at screening
5. On NRTI therapy against HBV for at least 12 weeks prior to day 1 or have HBV DNA < 10 IU/ml at screening, currently on locally approved NRTI therapy

Exclusion Criteria:

1. Serum ALT ≥ 5 × ULN
2. Any clinically significant chronic or acute medical or psychiatric condition that makes the participant unsuitable for participation.
3. History of significant liver disease from non-HBV or non-HDV etiology
4. History of allergic reactions, hypersensitivity, or intolerance to study drug, its metabolites, or excipients.
5. History of anaphylaxis
6. History of immune complex disease
7. History of autoimmune disorder
8. Current therapy or therapy within 24 weeks of screening with an immunomodulatory agent, immune checkpoint inhibitors, immunosuppressants, cytotoxic or chemotherapeutic agent, or chronic systemic corticosteroids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
HDV RNA < Lower Limit of Quantification (LLOQ), Target not detected (TND) at Week 24 | Week 24
HDV RNA < Lower Limit of Quantification (LLOQ), Target not detected (TND) 24 weeks after end of treatment. | 24 Weeks after End of Treatment

SECONDARY OUTCOMES:
Incidence of Treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) through Week 24, Week 48, Week 96, Week 120, Week 144, Week 192, and Week 240 | Week 24, Week 48, Week 96, Week 120, Week 144, Week 192, and Week 240
HDV RNA < Lower Limit of Quantification (LLOQ), Target not detected (TND) at Week 48, Week 96, Week 120, Week 144, Week 192 and Week 240 | Week 48 , Week 96, Week 120, Week 144, Week 192 and Week 240
Change from baseline in ALT at Week 24, Week 48, Week 96, Week 120, Week 144, Week 192, and Week 240 | Week 24, Week 48, Week 96, Week 120, Week 144, Week 192, and Week 240

CONTACTS AND LOCATIONS:
Locations (24):
- France (11):
  - Investigative Site, Bobigny
  - Investigative Site, Clichy
  - Investigative Site, Créteil
  - Investigative Site, Le Chesnay
  - Investigative Site, Limoges
  - Investigative Site, Lyon
  - Investigative Site, Montpellier
  - Investigative Site, Pessac
  - Investigative Site, Rennes
  - Investigative Site, Toulouse
  - Investigative Site, Villejuif
- Germany (4):
  - Investigative Site, Berlin
  - Investigative Site, Essen
  - Investigative Site, Frankfurt am Main
  - Investigative Site, Hanover
- Investigative Site, Milan, Italy
- Romania (2):
  - Investigative Site, Bucharest
  - Investigative Site, Craiova
- Spain (3):
  - Investigative Site, Barcelona
  - Investigative Site, Madrid
  - Investigative Site, Santander
- United Kingdom (3):
  - Investigative Site, London
  - Investigative Site, Manchester
  - Investigative Site, Nottingham